CLINICAL TRIAL: NCT00658580
Title: A Phase III Randomized Study Comparing A Chemotherapy With Cisplatin And Etoposide To A Etoposide Regimen Without Cisplatin For Patients With Extensive Small-Cell Lung Cancer
Brief Title: Randomized Study of Cisplatin-Etoposide Versus an Etoposide Regimen Without Cisplatin in Extensive Small-Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELCWP 01994
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Small Cell Lung Carcinoma, Extensive Disease
Keywords: Small cell lung carcinoma; Chemotherapy; Phase III randomised study
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PE regimen; Epirubicin; Ifosfamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Every 3 weeks intravenous cisplatin plus etoposide
  Interventions: Drug: Cisplatin + etoposide
- B (Experimental): Every 3 weeks intravenous epirubicin plus ifosfamide plus etoposide
  Interventions: Drug: Epirubicin + ifosfamide + etoposide

INTERVENTIONS:
Drug: Cisplatin + etoposide — Cisplatin 90 mg/m² day 1, every 3 weeks
  Etoposide 100 mg/m² days 1-3, every 3 weeks
  Arms: A
Drug: Epirubicin + ifosfamide + etoposide — Epirubicin 60 mg/m² day 1, every 3 weeks
  Ifosfamide (+ uromitexan) 1.5 g/m² days 1-3, every 3 weeks
  Etoposide 100 mg/m² days 1-3, every 3 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine if a cisplatin-etoposide regimen improves survival in comparison to a regimen containing etoposide and without platinum derivative.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of small-cell lung cancer
* Extensive disease (i.e. a disease with distant metastases or that cannot be included in a single irradiation field incorporating primary tumour, mediastinum and supraclavicular lymph node(s))
* Availability for participating in the detailed follow-up of the protocol
* Presence of an evaluable or measurable lesion
* Informed consent

Exclusion Criteria:

* Prior treatment with chemotherapy, radiotherapy or surgery
* Performance status < 60 on the Karnofsky scale
* A history of prior malignant tumor, except non-melanoma skin cancer or in situ carcinoma of the cervix or a cured cancer (defined as a disease-free interval > 5 years)
* White blood cells < 4000/mm3
* Platelets < 100000/mm3
* Serum bilirubin > 1.5 mg/100 ml
* Serum creatinine > 1.3 mg/100 ml and creatinine clearance <60 ml/min
* Recent myocardial infarction (less than 3 months prior to date of diagnosis)
* Congestive cardiac failure or cardiac arrhythmia uncontrolled by medical treatment
* Uncontrolled infectious disease
* Serious medical or psychological factors which may prevent adherence to the treatment schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2000-04; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Survival | Survival will be dated from the day of randomisation until death or last follow up

SECONDARY OUTCOMES:
Response rate | Every 3 cycles of chemotherapy
Toxicity | After every cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Sculier, MD, PhD, Study Chair — European Lung Cancer Working Party
Locations (4):
- Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels, Belgium
- Department of Pneumology CHRU Lille, Lille, France
- Hellenic Cancer Institute - St Savas Oncology Hospital, Athens, Greece
- Medical Oncology Hospital de Sagunto, Valencia, Spain

REFERENCES:
- [Derived] Berghmans T, Scherpereel A, Meert AP, Giner V, Lecomte J, Lafitte JJ, Leclercq N, Paesmans M, Sculier JP; European Lung Cancer Working Party (ELCWP). A Phase III Randomized Study Comparing a Chemotherapy with Cisplatin and Etoposide to a Etoposide Regimen without Cisplatin for Patients with Extensive Small-Cell Lung Cancer. Front Oncol. 2017 Sep 19;7:217. doi: 10.3389/fonc.2017.00217. eCollection 2017. PMID 28975084
- See also: Click here for more information on the protocol — http://www.elcwp.org
- See also: Trials registry of the French National Cancer Institute — http://www.e-cancer.fr